CLINICAL TRIAL: NCT03909490
Title: Does the Use of a Preference Elicitation Tool at Point of Care in Trigger Finger Change Decisional Conflict?
Brief Title: Trigger Finger Preference Elicitation Tool
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Logistics (research personnel)
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Robin Kamal, Assistant Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 45990
Record Dates: First submitted 2019-04-08; First posted 2019-04-10 (Actual); Last update posted 2021-11-12 (Actual); Status verified 2021-11

CONDITIONS: Trigger Finger; Trigger Thumb; Trigger Digit; Trigger Finger Disorder; Trigger Thumb, Left Thumb; Trigger Thumb, Right Thumb; Trigger Finger, Ring Finger; Trigger Finger, Index Finger; Trigger Finger, Middle Finger; Trigger Finger, Little Finger; Trigger Thumb, Unspecified Thumb; Trigger Finger, Unspecified Finger
MeSH Terms: conditions — Trigger Finger Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator)
  Interventions: Other: handout
- intervention- tool (Experimental)
  Interventions: Other: Preference elicitation tool

INTERVENTIONS:
Other: Preference elicitation tool — Ranking tool to assess patient preferences for trigger finger treatment
  Arms: intervention- tool
Other: handout — handout with information about trigger fingers
  Arms: Control

SUMMARY:
The purpose of this study is to evaluate a patient's level of decisional conflict for their treatment decision regarding their trigger finger, and study if the use of a preference elicitation tool at point of care is able to alter the level of decisional conflict

DETAILED DESCRIPTION:
All patients presenting to the Hand Surgery clinic for evaluation of a new trigger finger will be approached for inclusion in the study. Upon diagnosis, a patient diagnosed with a trigger will be informed of the study, asked if they would like to participate, and consented into the study. Patients will then be randomized to a control group versus our test group. The control group will be given a generic handout about trigger finger and the treatment options. They will then complete the decisional conflict survey without using the tool. The second group will use the tool and then complete the decisional conflict survey.

The standard of care is not being altered- all treatment options will still be available to patients and they have select whatever option is most in line with their preference for treatment. The purpose of the tool is to facilitate preference elicitation for treatment.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of trigger finger

Exclusion Criteria:

* prior trigger finger treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-03-20 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Decisional Conflict Scale (DCS) | Immediately after visit
  Decisional Conflict Scale (DCS) is a validated tool that measures a state of uncertainty about a course of action. DCS is a 16 item scale, scores range from 0-100, with higher scores indicating greater decisional conflict

CONTACTS AND LOCATIONS:
Overall Officials: Robin Kamal, Principal Investigator — Stanford University
Locations (1):
- Stanford Health Care, Redwood City, California, United States

IPD SHARING:
Plan to Share IPD: No